CLINICAL TRIAL: NCT03127592
Title: Phase III Randomized, Unicentric, Double-masked, Parallel Trial for the Efficacy and Tolerability of the Fixed Dose Combination of Etodolac 400 mg and Cyclobenzaprine 10 mg Versus the Isolated Active Substances (Flancox® 400 mg And Miosan® 10 mg) in Postoperative Pain Control After Impacted Third Molar Extraction
Brief Title: Phase III Efficacy and Tolerability Trial of the Fixed Dose Combination of Etodolac 400 mg and Cyclobenzaprine 10 mg Versus Isolated Active Substances in Pain Control After Impacted Third Molar Extraction
Acronym: FDCETCB-III
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: recruitment difficulty
Sponsor: Apsen Farmaceutica S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ETCAPS0317OR-III
Record Dates: First submitted 2017-04-17; First posted 2017-04-25 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain | interventions — Etodolac; cyclobenzaprine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): 1 active treatment (Fixed Dose Combination) + 2 placebos
  Interventions: Drug: Fixed Dose Combination
- Group 2 (Active Comparator): 1 active treatment (Cyclobenzaprine) + 2 placebos
  Interventions: Drug: Cyclobenzaprine
- Group 3 (Active Comparator): 1 active treatment (Etodolac) + 2 placebos
  Interventions: Drug: Etodolac

INTERVENTIONS:
Drug: Fixed Dose Combination — Fixed Dose Combination of Etodolac 400 mg + Cyclobenzaprine 10 mg
  Arms: Group 1
Drug: Etodolac — Individual drug
  Other Names: Flancox
  Arms: Group 3
Drug: Cyclobenzaprine — Individual drug
  Other Names: Miosan
  Arms: Group 2

SUMMARY:
This Phase III study will compare the efficacy and tolerability of a Fixed Dose Combination of Etodolac + Cyclobenzaprine versus the isolated drugs in postoperative pain control after impacted third molar extraction.

ELIGIBILITY:
Inclusion Criteria:

* Healthy research participants of both sexes (male and female non-pregnant), aged 18 years or over, underwent impacted third molar extraction surgery

Exclusion Criteria:

* Presence of any event and / or pathology at the site of interest that may interfere with and contraindicate the performance of the surgical procedure at the discretion of the Investigator, including periodontitis, odontogenic tumors or cysts (associated or not with the third molar), trauma, presence of Inflammation and / or infection;
* Present or past history of any cardiac, gastrointestinal, respiratory, hepatic, renal, endocrine, neurological, metabolic, psychiatric, hematological event;
* Previous diagnosis of alcohol and drug abuse defined by DSM-V;
* Current or past history (for less than 12 months) of smoking;
* Use of illicit drugs;
* History of bleeding / bleeding or coagulation disorders, gastric ulcer and / or active peptic hemorrhage;
* Any finding of clinical (clinical / physical), laboratory or cardiac evaluation (ECG) observation that is interpreted by the investigating physician as a risk to the participant;
* Use of drugs that potentially interfere with the kinetics / dynamics of acetaminophen or any other medicinal product considered clinically significant by the Investigator;
* Known hypersensitivity to the active principles used during the study (etodolac and cyclobenzaprine);
* Women in gestation or breastfeeding, as well as women who present a positive pregnancy test (β - hCG) during the study screening / selection period;
* Professionals directly involved in the realization of the present study and their relatives;
* Participant of the research that has participated in clinical study protocols in the last 12 (twelve) months, unless the Investigator deems that there may be direct benefit to it.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Superiority of the Fixed Dose Combination versus Isolated active substances | 4 hours
  The Primary outcome will be accessed by the individual response rate in relation to the pain intensity calculated by the Visual Analogic Scale (VAS) scale performed after 4 hours of administration of the first dose of medicines

SECONDARY OUTCOMES:
Individual response rate | 6h, 12h, 24h, 48h and 72h
  Individual response rate in relation to the evaluation of pain intensity calculated through the Visual Analogic Scale (VAS) measure in times 6h, 12h, 24h, 48h and 72h
Edema | 4 hours
  Absence of edema after 4 hours of drug administration and at the end of treatment
Mandibula constriction | 4 hours
  Absence of mandibular constriction after 4 hours of drug administration and at the end of treatment
Use of rescue medication | 3 days
  Proportion of participants requiring the use of rescue medication over the 3 days of treatment in each treatment group

CONTACTS AND LOCATIONS:
Locations (1):
- Azidus Brasil Pesquisa Científica e Desenvolvimento Ltda., Valinhos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No